CLINICAL TRIAL: NCT03830034
Title: Amino Acid Chelated Iron Versus Ferrous Fumarate in the Treatment of Iron Deficiency Anemia With Pregnancy: Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Shafy El Shahawy, lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IDA
Record Dates: First submitted 2019-02-02; First posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferrous fumarate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amino Acid chelated iron tab 15 mg group (Experimental): Contain 75 pregnant women will recommended to take ferrotrone(iron chelated amino acid containing 15mg elemental iron) prepared by egyptian pharmaceutical company (nerhadou) once daily (a dose recommended by the company of the product).
  Interventions: Drug: Amino Acid chelated iron tab 15 mg
- Ferrous Fumarate tab 350 mg( 115 mg elemental iron) group (Active Comparator): Contain 75 pregnant women will recommended to take ferrous fumarate e.g. Hema-caps (ferrous fumarate 350 mg with elemental iron 115mg) prepared by another egyptian pharmaceutical company (Amoun pharmaceutical company) once daily but in sever cases of iron deficiency anemia (Hb<9g/dl) this dose can be doubled as recommended by the company of the product.
  Interventions: Drug: Ferrous Fumarate tab 350 mg( 115 mg elemental iron)

INTERVENTIONS:
Drug: Amino Acid chelated iron tab 15 mg — Contain 75 pregnant women will recommended to take ferrotrone(iron chelated amino acid containing 15mg elemental iron) a dose recommended by the company of the product.
  Iron tablets should be taken at night or at least 1 hour prior to food to maximise absorption.
  Substances that inhibit absorption such as tannins & milk should be avoided but fruit juice contain ascorbic acid taken in conjunction with iron supplements increases their absorption.
  Follow up will be done for all the pregnant women included in our studies at baseline & then 4, 8 & 12 weeks after treatment at each visit breif history for outcomes and adverse effects will reviewed.
  Other Names: Ferrotron
  Arms: Amino Acid chelated iron tab 15 mg group
Drug: Ferrous Fumarate tab 350 mg( 115 mg elemental iron) — 75 pregnant women will recommended to take ferrous fumarate e.g. Hema-caps (ferrous fumarate 350 mg with elemental iron 115mg) prepared by another egyptian pharmaceutical company (Amoun pharmaceutical company) once daily but in sever cases of iron deficiency anemia (Hb<9g/dl) this dose can be doubled as recommended by the company of the product.
  Some instructions will be given to all the pregnant women included in our study as follow: Iron tablets should be taken at night or at least 1 hour prior to food to maximise absorption.
  Substances that inhibit absorption such as tannins & milk should be avoided but fruit juice contain ascorbic acid taken in conjunction with iron supplements increases their absorption.
  Follow up will be done for all the pregnant women included in our studies at baseline & then 4, 8 & 12 weeks after treatment at each visit breif history for outcomes and adverse effects will reviewed.
  Other Names: Haemacaps
  Arms: Ferrous Fumarate tab 350 mg( 115 mg elemental iron) group

SUMMARY:
Anemia is the commonest hematological disorder that occurs in pregnancy. According to the recent standard laid down by 'WHO', anemia is present when the Hemoglobin (Hb) concentration in the peripheral blood is 11 gm/dl or less. The most common cause of anemia in pregnancy is lack of iron. This study is done to compare the efficacy and tolerability of iron amino acid chelate and that of iron salts (ferrous fumarat).

DETAILED DESCRIPTION:
Anemia is the commonest hematological disorder that occurs in pregnancy. According to the recent standard laid down by 'WHO', anemia is present when the Hemoglobin (Hb) concentration in the peripheral blood is 11 gm/dl or less. The most common cause of anemia in pregnancy is lack of iron. This study is done to compare the efficacy and tolerability of iron amino acid chelate and that of iron salts (ferrous fumarat).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at 14 -18 weeks of gestation calculated from the first day of their last menstrual period and confirmed or modified by ultrasound
* Hemoglobin level 8-10.5 g/dL
* Serum ferritin<15µg/L

Exclusion Criteria:

* The presence of anemia from causes other than iron deficiency(e.g: Folat deficiency anemia,Vitamin B12 deficiency, ect…).
* Multiple gestations
* The presence of clinical and/or laboratory evidence of hepatic, renal, hematological or cardiovascular disease
* Patients with known gastritis
* History of mal-absorption syndrome
* Those with known hypersensitivity to iron preparations
* Those under current iron supplementation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — this trial conducted on treatment of iron deficiency anemia in pregnant women
Enrollment: 150 (Estimated)
Dates: Start 2019-02-02 (Actual); Primary Completion 2019-10-15 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobine (Hb) Rise | after 12 weeks of treatment.
  follow up CBC after 12 weeks of treatment given

SECONDARY OUTCOMES:
Hemoglobine (Hb) Rise | after 4,8 weeks of treatment.
  Follow up CBC after 4,8 weeks of treatment given
Adverse effects of the medication given | 3months
  constipation, nausea, allergy.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshahawy, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain shams university maternity hospital, Cairo, Egypt